CLINICAL TRIAL: NCT03846362
Title: A Prospective Multicenter Clinical Trial of Treatment Strategy Based on MRD Level After 2 Initial Courses of Chemotherapy in Children and Young Adults With Acute Myeloid Leukemia
Brief Title: A Prospective Multicenter Clinical Trial of MRD-based Treatment Strategy in Children and Young Adults With AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Collaborators: Physicians, Innovations, Science for Children Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2018-05
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia, Childhood
Keywords: AML; MRD; stem cell transplantation; pediatric; leukemia; haploidentical; TcRab-depletion; young adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intermediate risk MRD2>0,1% (Experimental): MRD2>0,1% - FLA - MRD3 - HSCT
  Interventions: Other: HSCT

INTERVENTIONS:
Other: HSCT — allogenic HSCT from 5-8 HLA-MM family donor as a first choice for patients with initial high risk of relapse and for patients with MRD2>0,1% and initial intermediate risk

SUMMARY:
Minimal-residual disease (MRD) will be measured either by flow cytometry, or polymerase chain reaction (PCR) methods, in 3 check-points and it will be one of the decision-making control parameter for the optimal therapy tactics.

Patients with initially high-risk group and those with high MRD after 2 initial courses of chemotherapy will be assigned to the allogenic transplantation of the hematopoietic stem cells from Human Leucocyte Antigen (HLA) matched or haploidentical family donors.

DETAILED DESCRIPTION:
Genetic alterations in acute myeloid leukemia (AML) clone are well known prognostic risk factors of AML relapse. Standard risk group includes favorable t (15;17) (q22; q21) and inv (16)/t (16;16). High-risk patients have a complex karyotype rearrangement (3 and more), inversion of the long arm in 3rd chromosome and EVI1 gene rearrangement, monosomy 5 and 7, translocations involving KMT2A gene and several rare translocations. All other genotype alterations attributed to the moderate risk group.

Besides genetic factors, detection of the minimal residual disease (MRD) after initial chemotherapy and its decrease rate after 1st postremission chemotherapy with high dose Cytarabine and anthracyclines, plays a crucial role in the development of the morphologic relapse. Patients with PCR-MRD<0,1% after 2 courses of chemotherapy have a 30% or less risk of relapse, while PCR-MRD>0,1% - over 70%. In the clinical trial investigators are planning to measure MRD either by immune-phenotype, or PCR methods, in 3 check-points and it will be one of decision-making control parameter for the optimal therapy tactics.

Patients with initially high-risk group and those with high MRD after 2 initial courses of chemotherapy will be assigned to the allogenic transplantation of the hematopoietic stem cells from HLA- matched or haploidentical family donors.

ELIGIBILITY:
Inclusion Criteria:

1. de novo acute myeloid leukemia
2. signed informed consent

Exclusion Criteria:

diagnosis of: Fanconi anemia, acute promyelocytic leukemia, MDS, JMML, AML as secondary malignancy, Dawn syndrome.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival (RFS) | 1 year
  relapse-free survival from date of diagnosis till date of relapse, or date of death (whichever comes first) or date of last follow up

SECONDARY OUTCOMES:
overall survival (OS) | 1 year
event-free survival (EFS) | 2 years
  Event=relapse/nonresponse, death or second malignancy
The proportion of of patients with severe adverse effects | 6 months
  The proportion of of patients with severe adverse effects of therapy according to CTCAE (ver 4.3)
The proportion of of patients with severe infections | 1 month
  The proportion of of patients with severe infections: number of episodes, grade, after each course of chemotherapy
The proportion of of patients with severe cardiotoxicity | 1 year
  The proportion of of patients with severe cardiotoxicity: number of episodes and %EF by echocardiogam
MRD dynamic | 1 months
  MRD (IFT and/or PCR) dynamic between check-points
MRD specificity and sensitivity | 1, 2, 3 months
  MRD specificity and sensitivity in relapse prognosis
Cumulative incidence of relapse | 6 months, 1 year
  competing event - death in CR
Cumulative incidence of transplant-related mortality | 6 months after HSCT
  for transplanted patients
Cumulative incidence of aGvHD II-IV grade | 100 days after HSCT
  for transplanted patients
Cumulative incidence of cGvHD | 1 year after HSCT
  for transplanted patients

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Maschan, Principal Investigator — National Research Center for Pediatric Hematology , Moscow, Russian Federation; Michael Maschan, Study Director — National Research Center for Pediatric Hematology , Moscow, Russian Federation; Galina Novichkova, Study Chair — National Research Center for Pediatric Hematology , Moscow, Russian Federation
Locations (2):
- Russia (2):
  - Regional Children's Clinical Hospital № 1, Yekaterinburg, Sverdlovsk Oblast
  - Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow